CLINICAL TRIAL: NCT01746563
Title: Intravitreal Ranibizumab Combined With Panretinal Photocoagulation in Patients With Treatment-Naive Proliferative Diabetic Retinopathy
Brief Title: Intravitreal Ranibizumab Combined With Panretinal Photocoagulation in Patients With Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Araujo Ferraz, Ophthalmologist, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: USP-RBZ2012
Record Dates: First submitted 2012-12-06; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Diabetic Retinopathy; Retinal Diseases; Eye Diseases; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases
Keywords: Proliferative Diabetic Retinopathy; Ranibizumab; Panretinal Photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Diseases; Eye Diseases; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases | interventions — Ranibizumab; lactitol; Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Experimental): Ranibizumab 0,05 mg intravitreal injection
  Interventions: Drug: Ranibizumab; Procedure: Laser therapy
- Laser Therapy (Active Comparator): Laser Therapy alone
  Interventions: Procedure: Laser therapy

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection
  Other Names: Lucentis (Novartis)
  Arms: Ranibizumab
Procedure: Laser therapy — Laser therapy

SUMMARY:
To evaluate the efficacy of combination therapy with ranibizumab (RBZ) and panretinal photocoagulation (PRP) versus PRP alone in patients with treatment-naive bilateral proliferative diabetic retinopathy (PDR) as measured by mean change in visual acuity (VA), mean change in central retinal thickness (CRT) as measured by time-domain optic coherence tomography (TD-OCT) and incidence of vitreous hemorrhage (VH).

DETAILED DESCRIPTION:
Comparative efficacy of combined treatment including intravitreal injection of 0.5 mg of Lucentis (ranibizumab) and laser photocoagulation for patients with Proliferative Diabetic Retinopathy (PDR).

Objectives:

Primary objective:

The primary objective will be to evaluate the efficacy of combined treatment with ranibizumab and laser photocoagulation versus laser photocoagulation alone in patients with severe PDR by the mean change in BCVA at V7/M6 compared to baseline. The Best Visual Acuity (BCVA) measured by the Early Treatment Diabetic Retinopathy Study (EDTRS).

Secondary objectives:

To evaluate differences in Optic Coherence Tomography (OCT) retinal thickness and total macular volume of combined treatment regiment including intravitreal injection of 0,5 mg of Lucentis (ranibizumab) and laser photocoagulation for patients with PDR at visit 7 compared to the baseline assessments.

To evaluate the percentage of patients that present with vitreous hemorrhage after the beginning of the laser treatment at visit 7 compared to the baseline assessments.

Strategic goal:

The main goal of this study is to evaluate if the use of intravitreal ranibizumab in eyes submitted to Pan-Retinal Photocoagulation (PRP) due to PDR induces less macular edema and less vitreous hemorrhage and therefore leads to a better visual outcome

ELIGIBILITY:
Inclusion Criteria:

* Naive Proliferative diabetic retinopathy eyes.
* Best Corrected-Visual Acuity at baseline > 20/320 in the study eye
* Patients with and without diabetic macular edema
* Type II diabetic subjects as defined by the World Health Organization aged ≥ 18 years.
* Women must be using effective contraception
* Ability to provide written informed consent.
* Indication of panretinal photocoagulation in both eyes

Exclusion Criteria:

* Vitreous hemorrhage or pre-retinal hemorrhage
* Eyes with prior scatter (panretinal) or focal/grid photocoagulation, within the previous 6 months
* Atrophy/scarring/fibrosis/ hard exudates involving the center of the macula.
* Cataract
* Any intraocular surgery within 6 months before trial enrollment
* Previous vitrectomy.
* Any of the following underlying systemic diseases:
* History or evidence of severe cardiac disease or previous thrombus-embolic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Macular Evaluation | 6 Months
  Changes between visual acuity from baseline to month 6.

SECONDARY OUTCOMES:
Structural Macular Evaluation | 06 months
  Change on retinal thickness between baseline and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Walter Y Takahashi, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Rentiya ZS, Ferraz DA, Hutnik R, Bae J, Machado CG, Mucciolli C, Motta AALD, Ribeiro LZ, Guan Z, Preti RC, Takahashi WY. Evaluation of contrast sensitivity in non-high-risk proliferative diabetic retinopathy treated with panretinal photocoagulation with and without intravitreal injections of ranibizumab. Arq Bras Oftalmol. 2022 Jan-Feb;85(1):37-45. doi: 10.5935/0004-2749.20220006. PMID 34586227
- [Derived] Ferraz DA, Vasquez LM, Preti RC, Motta A, Sophie R, Bittencourt MG, Sepah YJ, Monteiro ML, Nguyen QD, Takahashi WY. A randomized controlled trial of panretinal photocoagulation with and without intravitreal ranibizumab in treatment-naive eyes with non-high-risk proliferative diabetic retinopathy. Retina. 2015 Feb;35(2):280-7. doi: 10.1097/IAE.0000000000000363. PMID 25272318